CLINICAL TRIAL: NCT01801124
Title: Evaluation of the Safety and Efficacy of EXPAREL® When Infiltrated Into the Transversus Abdominis Plane (TAP) for Prolonged Postoperative Analgesia in Subjects Undergoing Unilateral Abdominal Hernia Repair
Brief Title: EXPAREL Infiltrated Into the TAP for Postoperative Analgesia in Unilateral Abdominal Hernia Repair
Acronym: 702
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA402S23B702
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Results first posted 2013-09-11 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Hernia
Keywords: analgesia; hernia repair
MeSH Terms: conditions — Hernia; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EXPAREL (Experimental): undiluted EXPAREL 266 mg
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: EXPAREL — single dose 266 mg of undiluted EXPAREL
  Other Names: bupivacaine liposome injectable suspension

SUMMARY:
Phase 4 study evaluating the effectiveness of EXPAREL when infiltrated into the the Transversus Abdominis Plane (TAP).

DETAILED DESCRIPTION:
This is a prospective, open-label, non-randomized study evaluating the effectiveness of abdominal analgesia when using 266 mg EXPAREL to infiltrate into the TAP unilaterally.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 18-75 years inclusive, and ASA physical status 1-3.
* Undergoing open repair of a unilateral abdominal hernia below the level of the umbilicus.
* Abdominal incision length of 3-12 cm.
* Subjects must be physically and mentally able to participate in the study and complete all study assessments.
* Subjects must be able to give fully informed consent to participate in this study after demonstrating a good understanding of the risks and benefits of the proposed components of the TAP infiltration.

Exclusion Criteria:

* History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics
* Any subject whose anatomy, or surgical procedure, in the opinion of the Investigator, might preclude the potential successful performance of a TAP infiltration.
* Any subject who in the opinion of the Investigator, might be harmed or be a poor candidate for participation in the study.
* Any subject, who in the opinion of the Investigator, is on chronic pain medicine.
* Any female subject who is currently pregnant.
* Subjects who have received any investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during their participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kronenfeld, MD, Principal Investigator — Maimonides
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 20 July 2012 and 27 November 2012 at one site in the USA.
Pre-assignment Details: Subjects were not excluded.
Groups:
- EXPAREL: All subjects received a total of 266mg EXPAREL (bupicavaine liposome injectable suspension) diluted with preservative-free 0.9% normal saline to a volume of 30mL. Study drug was to be administered with ultrasound guidance by injection through a needle or catheter into the tissue plane between the transversus abdominis and internal oblique muscles of the abdominal wall.
Period: Overall Study
Arm/Group | EXPAREL
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EXPAREL
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Postsurgical Analgesic Use
Description: The effectiveness of abdominal analgesia from the infiltration into the TAP as measured by the subject's overall postsurgical analgesic use in morphine equivalents (mg)
Time Frame: 10 days
Population: The analysis population comprised all enrolled subjects.
Measure: Mean (Standard Deviation); unit: mg (morphine equivalents)
Groups:
- EXPAREL: Subjects receiving 266 mg EXPAREL to infiltrate into the bilateral TAPs.
Arm/Group | EXPAREL
Number analyzed (Participants) | 13
mg (morphine equivalents) | 9.7 (17.41)

2. Secondary Outcome: Postsurgical AEs and SAEs Through Day 30.
Description: Adverse events and serious adverse events through Day 30 will be examined in order to assess the safety of EXPAREL.
Time Frame: 30 days
Population: The analysis population comprised all enrolled subjects.
Measure: Number; unit: AEs
Arm/Group | EXPAREL
Number analyzed (Participants) | 13
AEs | 0

ADVERSE EVENTS:
Time Frame: Through Day 30
Description: Adverse events were collected by the investigator from the time of signing the informed consent form through 30 days post surgery.
Arm/Group | EXPAREL
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No